CLINICAL TRIAL: NCT06841744
Title: Effects of Diaphragmatic Breathing on Pain, Function, Balance and Quality of Life in Pregnant Women With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Kübra Akkurt, Physiotherapist, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0196
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Breathing Group (Experimental)
  Interventions: Other: Diaphragmatic Breathing Exercise; Other: Information brochure
- Control Group (Active Comparator)
  Interventions: Other: Information brochure

INTERVENTIONS:
Other: Diaphragmatic Breathing Exercise — Diaphragmatic breathing exercises will be performed twice a day, completing 3 sets of 10 repetitions, 5 days a week for 6 weeks, as instructed by the researcher physiotherapist.
  Arms: Diaphragmatic Breathing Group
Other: Information brochure — An information brochure on ergonomic strategies for managing low back pain during pregnancy will be provided.

SUMMARY:
The aim of the study was to investigate the effects of diaphragmatic breathing on pain, function, balance and quality of life in pregnant women with low back pain.

DETAILED DESCRIPTION:
Individuals with pregnancy-related low back pain who present to the Obstetrics and Gynecology Clinic of İzmir Menemen State Hospital are identified as the study population. Patients meeting the eligibility criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Pregnancy between 19-29 weeks
* Low back pain that started with pregnancy (at least 1 week; no previous history of low back pain)
* No treatment for the lumbar region or spine in the last 3 months

Exclusion Criteria:

* History of cardiovascular disease
* Multiple pregnancy
* Medical complications (e.g., bleeding, pre-eclampsia, placenta previa, etc.)
* Diagnosed cognitive disorders
* High-risk pregnancy
* History of abdominal and/or thoracic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, 6 weeks
  The Numeric Pain Rating Scale (NPRS) assesses pain severity using a 0-10 scale, where 0 represents "no pain" and 10 represents "the worst pain imaginable."
Oswestry Disability Index | Baseline, 6 weeks
  A questionnaire measuring disability associated with low back pain.

SECONDARY OUTCOMES:
Timed up and go test | Baseline, 6 weeks
  It measures the time required for a person to rise from a chair, walk three meters, turn, walk back to the chair, and sit down.
The Single Leg Stance Test | Baseline, 6 weeks
  The Single Leg Stand Test will be performed on the dominant leg, with eyes open and closed.
Quality of Life in Pregnancy Scale | Baseline, 6 weeks
  The Quality of Life in Pregnancy Scale aims to assess the quality of life of women with a normal pregnancy and consists of 9 items.The total score of the scale ranges from 9 to 45, with lower scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Izmir, Çigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No